CLINICAL TRIAL: NCT06874829
Title: Post-activation Performance Enhancement in Multi- vs Single-Joint Movements: A Comparative Study of BFR and EMS in Male Volleyball Athletes
Brief Title: Post-Activation Performance Enhancement in Single and Multi-Joint Exercises With BFR and EMS in Male Volleyball Players
Acronym: PAPE-BFR-EMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Neslihan AKÇAY, Assoc. Prof. Dr., Karabuk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UKarabuk-2
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Volleyball Players; Post Activation Potentiation; Muscle Strength
Keywords: Post-activation performance; Blood Flow Restriction Exercise; volleyball; Hand Grip Strength; Service Speed
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same is true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Blood flow restriction (Active Comparator): In the BFR group, 50% of the arterial occlusion pressure (AOP) was used.Bench press (multi-joint) and triceps push-down (single-joint) exercises were used in the conditions.
  Interventions: Other: Blood Flow Restriction
- Electrical muscle stimulation (Active Comparator): In the EMS group, a 75 Hz current was applied. Bench press (multi-joint) and triceps push-down (single-joint) exercises were used in the conditions.
  Interventions: Other: Electrical Muscle Stimulation
- Low Load Resistance Exercise (Active Comparator): In the Low Resistance Exercise group, only exercise was performed without any condition (BFR or EMS. Bench press (multi-joint) and triceps push-down (single-joint) exercises were used in the conditions.
  Interventions: Other: Low-Load Resistance Exercise

INTERVENTIONS:
Other: Electrical Muscle Stimulation — EMS will be applied bilaterally to the wrist flexor and elbow extensor muscles using a portable EMS stimulator (Compex Rehab 400, Medicompex SA, Ecublens, Switzerland). Four 2 mm thick, self-adhesive electrodes (5x5 cm) will be placed on the superficial aspect of each muscle group. The athletes will simultaneously receive EMS intervention with a pulse frequency of 75 Hz and a duration of 400 μs (19 seconds rest between pulses) during bench press and triceps pushdown exercises. Bench press and triceps push down exercises will be performed with 30% 1TM, 30-15-15-15 repetitions and thirty seconds rest between sets.
  Other Names: EMS
  Arms: Electrical muscle stimulation
Other: Blood Flow Restriction — The arterial occlusion pressures (AOP) of the athletes randomized to the experimental group will be obtained automatically with the digital LED display CAC device BFR Unit (Fit Cuffs BFR Unit, Denmark). The AOP pressure device BFR Unit (Fit Cuffs BFR Unit, Denmark) will be used to apply 50% occlusion pressure during exercise. Bench press and triceps push down exercises will be performed with 30% 1TM, 30-15-15-15 repetitions and thirty seconds rest between sets.
  Other Names: BFR
  Arms: Blood flow restriction
Other: Low-Load Resistance Exercise — Bench press and triceps pushdown exercises will be performed with 30% 1RM, 30-15-15-15 repetitions and 30 seconds rest between sets.
  Other Names: LL-RE
  Arms: Low Load Resistance Exercise

SUMMARY:
Investigators used a randomized controlled crossover design to compare the effect of blood flow restriction (BFR) and electrical muscle stimulation (EMS) protocols on post-activation performance enhancement (PAPE) in multi-joint versus single-joint exercises. Participants took part in six test sessions 72 hours apart. In the BFR group, 50% of the arterial occlusion pressure (AOP) was used. In the EMS group, a 75 Hz current was applied. In the Low Resistance exercise group, only exercise was performed without any condition. Bench press (multi-joint) and triceps push-down (single-joint) exercises were used in the conditions.

DETAILED DESCRIPTION:
Participants took part in six test sessions 72 hours apart. All tests were performed between 2 and 4 pm to reduce the influence of circadian rhythms or fatigue on performance. Anthropometric measurements, 1 RM test, and grip strength and serving speed tests were determined before the practice session on the first day as a control condition. On the other six experimental days, players were randomly assigned to protocols (BFR, EMS, and LOW-LOAD) using software (http://www.randomizer.org). In the BFR group, 50% of the arterial occlusion pressure (AOP) was used. In the EMS group, a 75 Hz current was applied. In the Low Resistance exercise group, only exercise was performed without any condition. Bench press (multi-joint) and triceps push-down (single-joint) exercises were used in the conditions. In all protocols, participants performed a standardized warm-up protocol consisting of a 5-minute run at 9 km/h on a treadmill and a general warm-up consisting of 3 minutes of whole-body light stretching exercises. Following the warm-up and pre-exercise protocols, grip strength and service speed tests were performed with rest periods.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male volleyball athletes
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 18 years old
* Having a chronic disease
* Contraindication for Electromyostimulation (EMS)
* Contraindication for Blood Flow Restriction (BFR)
* Contraindications for exercise

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-08-09 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Service speed | From baseline to the end of treatment at 8 weeks
  Service speed will assess by standard radar apparatus (Net Playz Smart Pro Speed Radar, USA) and will record in km/h.
Hand Grip strength | From baseline to the end of treatment at 8 weeks
  Hand grip strength will assess by hand grip dynamometer (Takei 5,101, Tokyo, Japan) and will record in kg.

OTHER OUTCOMES:
Bench Press 1Repetition maximum Test | Baseline
  The 1RM values of the participants will assess by using a bench press machine.
Triceps Push Down 1 repetition maximum Test | Baseline
  The participants will instruct to assume a standing position in front of the triceps push-down machine, holding the bar with both hands in the pronated position at shoulder width. During the execution of this exercise, the participants will maintain their arms near their torso, ensuring that there was no contact between the arms and the body.
Anthropometric Measurements 1 | Baseline
  Participants' height (cm) will assess by using a stadiometer (Holtain Stadiometer, England).
Anthropometric Measurements 2 | Baseline
  Body weight (kg) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 3 | Baseline
  Body mass index (BMI) (kg/m2) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 4 | Baseline
  Body fat percentage (%) will asses by Inbody 270 (Biospace, California, USA).
  Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan AKCAY, Doctorate, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keskin K, Akcay N, Ozmen T, Contarli N, Yildiz KC, Sofuoglu C, Kamis O, Rolnick N, de Queiros VS, Montoye A. Effects of different pre-exercise strategies on jumping performance in female volleyball players. J Sports Med Phys Fitness. 2025 Jan;65(1):59-68. doi: 10.23736/S0022-4707.24.16196-8. Epub 2024 Oct 3. PMID 39360986